CLINICAL TRIAL: NCT06736587
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Dose, Dose-escalation Phase 1 Clinical Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DWP212525 in Healthy Male Volunteers
Brief Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase 1 Clinical Tiral in Healthy Male Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DW_DWP212525101
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort2 (Experimental): SAD
  Interventions: Drug: DWP212525 30mg; Drug: DWP212525 placebo
- Cohort3 (Experimental): SAD
  Interventions: Drug: DWP212525 50mg; Drug: DWP212525 placebo
- Cohort4 (Experimental): SAD
  Interventions: Drug: DWP212525 100mg; Drug: DWP212525 placebo
- Cohort5 (Experimental): SAD
  Interventions: Drug: DWP212525 200mg; Drug: DWP212525 placebo
- Cohort6 (Experimental): SAD
  Interventions: Drug: DWP212525 400mg; Drug: DWP212525 placebo
- Cohort7 (Experimental): MAD
  Interventions: Drug: DWP212525 30mg; Drug: DWP212525 placebo
- Cohort8 (Experimental): MAD
  Interventions: Drug: DWP212525 50mg; Drug: DWP212525 placebo
- Cohort9 (Experimental): MAD
  Interventions: Drug: DWP212525 100mg; Drug: DWP212525 placebo
- Cohort10 (Experimental): MAD
  Interventions: Drug: DWP212525 200mg; Drug: DWP212525 placebo
- Cohort1 (Experimental): SAD
  Interventions: Drug: DWP212525 10mg; Drug: DWP212525 placebo

INTERVENTIONS:
Drug: DWP212525 10mg — DWP212525 10mg
  Arms: Cohort1
Drug: DWP212525 30mg — DWP212525 30mg
  Arms: Cohort2; Cohort7
Drug: DWP212525 50mg — DWP212525 50mg
  Arms: Cohort3; Cohort8
Drug: DWP212525 100mg — DWP212525 100mg
  Arms: Cohort4; Cohort9
Drug: DWP212525 200mg — DWP212525 200mg
  Arms: Cohort10; Cohort5
Drug: DWP212525 400mg — DWP212525 400mg
  Arms: Cohort6
Drug: DWP212525 placebo — DWP212525 placebo

SUMMARY:
The safety and tolerability of single and multiple administration of DWP212525

DETAILED DESCRIPTION:
The safety and tolerability of single and multiple administration of DWP212525 will be evaluated in healthy adult male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers aged 19 to 55 years, Caucasian
2. Those with a body weight ≥ 50.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 kg/m2 to ≤ 30.0 kg/m2
3. Received a sufficient explanation on this study
4. Eligible as subjects in the study

Exclusion Criteria:

1. History of diseases such as clinically significant disease of hepatobiliary
2. Following conditions applicable to clinically significant acute or chronic infections or the past history confirmed via an interview
3. Hemato-oncologic diseases, including malignant tumor diagnosis
4. Past history of tuberculosis infection or confirmed tuberculosis in the IGRA test and chest X-ray test

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of DWP212525 and metabolite M16 | Day 1 0 hour (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72hours post-dose
  AUClast, AUCinf
Concentration of DWP212525 and metabolite M16 | Day 1 0 hour (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72hours post-dose
  Cmax
Concentration of DWP212525 and metabolite M16 | Day 1 0 hour (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72hours post-dose
  Tmax
Concentration of DWP212525 and metabolite M16 | Day 1 0 hour (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72hours post-dose
  t1/2
Concentration of DWP212525 and metabolite M16 | Day 1 0 hour (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72hours post-dose
  CL/F
Concentration of DWP212525 and metabolite M16 | Day 1 0 hour (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72hours post-dose
  Vz/F

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No